CLINICAL TRIAL: NCT01864681
Title: A Phase II, Randomized, Placebo Controlled Study to Evaluate the Efficacy of the Combination of Gefitinib and Metformin in Patients With Locally Advanced and Metastatic Non-Small-Cell-Lung-Cancer
Brief Title: Combination of Metformin With Gefitinib to Treat NSCLC
Acronym: CGMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yong He, Director of Department of Respiratory Diseases, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012XLC07
Record Dates: First submitted 2013-05-25; First posted 2013-05-29 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: NSCLC; EGFR Gene Amplification; Advanced Cancer; Stage IIIB NSCLC; Stage IV NSCLC
Keywords: NSCLC; TKIs; Metformin; PFS; overall survival; IL-6
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Gefitinib and metformin. Metformin starting at a dose of 500 mg twice a day, orally with meals. After one week, increase the dose of metformin to 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin treatment will be initiated one week before beginning TKI therapy, if possible, but TKI therapy will not be delayed for metformin loading.
  Interventions: Drug: Gefitinib and Metformin
- Arm B (Placebo Comparator): Gefitinib and placebo. Placebo was given to patients in the same way as that of metformin in Arm A.
  Interventions: Drug: Gefitinib and placebo

INTERVENTIONS:
Drug: Gefitinib and Metformin — Gefitinib will be administered once every day. If subject has complete response, partial response, stable disease, or unacceptable toxicity.
  Arms: Arm A
Drug: Gefitinib and placebo — Gefitinib will be administered once every day. If subject has complete response, partial response, stable disease, or unacceptable toxicity.
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine whether metformin in combination with gefitinib are effective in patients with previously untreated advanced or metastatic Non-Small-Cell Lung cancer with epidermal growth factor receptor (EGFR) mutations

DETAILED DESCRIPTION:
Primary Objectives: To determine the 1 year progression-free survival (PFS) of the combination of metformin and gefitinib in patients who harbors EGFR-mutant with previously untreated advanced or metastatic pulmonary adenocarcinoma.

Secondary Objectives:

A. To evaluate the response to therapy and overall survival of the combination of metformin with gefitinib in patients who harbors EGFR-mutant with previously untreated advanced or metastatic pulmonary adenocarcinoma.

B. To acquire preliminary data regarding the effects of metformin on interleukin-6 (IL-6) levels in tumor and serum.

Treatment will be administered on an outpatient basis. Metformin starting at a dose of 500 mg twice a day, orally with meals. After one week, increase the dose of metformin to 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin treatment will be initiated one week before beginning gefitinib, if possible, but gefitinib administration will not be delayed for metformin loading.

Gefitinib will be administered 250mg QD continuously. Metformin will be administered continuously, beginning one week before beginning gefitinib, if possible, but tyrosine kinase inhibitors (TKI) will not be delayed for metformin loading.

Maintenance Therapy Patients responding to this therapy will be maintained with metformin (1000 mg twice daily) and gefitinib.

Duration of Therapy

In the absence of treatment delays due to adverse events, treatment may continue until one of the following criteria applies:

1. Disease progression,
2. Intercurrent illness that prevents further administration of treatment,
3. Unacceptable adverse events(s),
4. Patient decides to withdraw from the study, or
5. General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Histologically or cytologically confirmed non small cell carcinoma of the lung who harbors EGFR-mutation and are previously untreated
* Patient must have measurable stage IV disease (includes M1a, M1b stages or recurrent disease) (according to the 7th edition of the tumor node metastasis (TNM) classification system). However, patients with T4NX disease (stage III B) with nodule(s) in ipsilateral lung lobe are not eligible, because such patients were not included in historical controls.
* Patients be age >18 years and < 75 years.
* Patients must have a Life Expectancy of greater than 12 weeks.
* Patients must have an electrocorticography (ECOG) performance status 0 or 1 (Karnofsky > 70%).
* Patients must have normal organ and marrow function as defined below, within one week prior to randomization:

absolute neutrophil count >1,500/mL platelets > 100,000/mL total bilirubin: within normal institutional limits AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal creatinine ≤ 1.5 X institutional upper limit of normal urine dipstick for proteinuria of < less than 1+. If urine dipstick is > 1+ then a 24 hour urine for protein must demonstrate < 500 mg of protein in 24 hours to allow participation in the study.

* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients must have an international normalized ratio (INR) < 1.5 and a partial thromboplastin time (PTT) no greater than upper limits of normal within 1 week prior to randomization.
* Patients with a history of hypertension must be well-controlled (<150 systolic/<100 diastolic) on a stable regimen of anti-hypertensive therapy.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
* Patients receiving chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory agents known to inhibit platelet function. Treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and/or cilostazol (Pletal)is also not allowed.
* Patients receiving therapeutic anticoagulation. Prophylactic anticoagulation of venous access devices is allowed provided Section 3.10 is met. Caution should be taken on treating patients with low dose heparin or low molecular weight heparin for DVT prophylaxis during treatment with bevacizumab as there may be an increased risk of bleeding.
* Prior use of chemotherapy.
* Patients receiving immunotherapy, hormonal-therapy and or radiotherapy within 2 weeks prior to entering the study. Note: Those who have not recovered from adverse events due to these agents administered will be considered ineligible.
* Patients receiving any other investigational agents.
* Patients with uncontrolled brain metastasis. Note: Patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin and paclitaxel or other agents used in the study are excluded.
* Women that are pregnant or breastfeeding Note: Pregnant women are excluded from this study because the agents used in this study may be teratogenic to a fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with paclitaxel, breastfeeding women are also excluded from this study.
* Patients that are HIV-positive on combination antiretroviral therapy due to the potential for lethal infections when treated with marrow-suppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
PFS | 1 year
  One year progression-free survival (PFS) of the patients.

SECONDARY OUTCOMES:
Response to therapy and overall survival | 2 years
  The response to therapy and overall survival of the patients.

OTHER OUTCOMES:
IL-6 level | 2 years
  IL-6 level in tumors and blood serum of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yong He, MD, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (1):
- Department of Respiratory Diseases, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Li KL, Li L, Zhang P, Kang J, Wang YB, Chen HY, He Y. A Multicenter Double-blind Phase II Study of Metformin With Gefitinib as First-line Therapy of Locally Advanced Non-Small-cell Lung Cancer. Clin Lung Cancer. 2017 May;18(3):340-343. doi: 10.1016/j.cllc.2016.12.003. Epub 2016 Dec 22. PMID 28065465